CLINICAL TRIAL: NCT00238121
Title: A Phase II Study of BAY 43-9006 in Advanced/Recurrent Uterine Carcinoma/Carcinosarcoma
Brief Title: Sorafenib in Treating Patients With Advanced or Recurrent Uterine Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00068; 13572A; CDR0000445181; N01CM62203 (NIH)
Record Dates: First submitted 2005-10-12; First posted 2005-10-13 (Estimated); Results first posted 2014-06-10 (Estimated); Last update posted 2015-11-20 (Estimated); Status verified 2014-01

CONDITIONS: Recurrent Uterine Sarcoma; Stage III Uterine Sarcoma; Stage IV Uterine Sarcoma; Uterine Carcinosarcoma
MeSH Terms: interventions — Sorafenib

ARMS (1):
- Treatment (Experimental): Patients receive oral sorafenib twice daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: sorafenib tosylate

INTERVENTIONS:
Drug: sorafenib tosylate — Given orally
  Other Names: BAY 43-9006; BAY 43-9006 Tosylate Salt; BAY 54-9085; Nexavar; SFN

SUMMARY:
Sorafenib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor. This phase II trial is studying how well sorafenib works in treating patients with advanced or recurrent uterine cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the objective response rate in patients with advanced or recurrent uterine cancer treated with sorafenib.

II. Determine the toxic effects of this drug in these patients.

SECONDARY OBJECTIVES:

I. Determine progression-free survival of patients treated with this drug.

OUTLINE: This is a multicenter study. Patients are stratified according to histology (carcinoma vs carcinosarcoma).

Patients receive oral sorafenib twice daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* No prior sorafenib
* Histologically or cytologically confirmed uterine carcinoma or carcinosarcoma:

  * Advanced or recurrent disease
  * Not amenable to curative surgery or radiotherapy
* Measurable disease:

  * At least 1 unidimensionally measurable lesion >= 20 mm by conventional techniques OR >= 10 mm by spiral CT scan
* Tumor tissue block must be available
* No known brain metastases
* Performance status:

  * ECOG 0-2 OR
  * Karnofsky 60-100%
* Hematopoietic:

  * Absolute neutrophil count >= 1,500/mm3
  * Platelet count >= 100,000/mm3
  * No bleeding diathesis
* Hepatic:

  * Bilirubin normal
  * AST and ALT =< 2.5 times upper limit of normal
* Renal:

  * Creatinine =< 1.5 mg/dL OR
  * Creatinine clearance >= 60 mL/min
* Cardiovascular:

  * No uncontrolled hypertension, defined by 1 of the following:

    * Blood pressure > 150/100 mm Hg
    * Currently taking > 1 antihypertensive agent
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No other active malignancy
* No history of allergic reactions attributed to compounds of similar chemical or biological composition to sorafenib
* No ongoing or active infection
* No psychiatric illness or social situation that would preclude study compliance
* No swallowing dysfunction that would preclude study drug ingestion
* No other uncontrolled illness
* Prior biological response modifier therapy allowed
* No prior antiangiogenesis therapy
* No prior MAPK-signaling agents
* No prior vascular endothelial growth factor receptor (VEGFR) inhibitors
* No more than 1 prior chemotherapy regimen
* More than 4 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin)
* Prior hormonal therapy allowed
* Prior radiotherapy allowed provided the only site of measurable disease was not located within the radiation port OR disease has progressed since completion of therapy
* Recovered from all prior therapy
* Concurrent warfarin allowed provided all of the following are true:

  * Patient is therapeutic on a stable warfarin dose
  * INR target range =< 3
  * Patient is monitored with weekly INR testing
  * No active bleeding or pathological condition that carries a high bleeding risk
* No concurrent combination antiretroviral therapy for HIV-positive patients
* No concurrent cytochrome P450 enzyme-inducing antiepileptic drugs (e.g., phenytoin, carbamazepine, or phenobarbital)
* No concurrent rifampin
* No concurrent Hypericum perforatum (St. John's wort)
* No other concurrent investigational agents
* No other concurrent anticancer therapy
* More than 4 weeks since prior radiotherapy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2005-02; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gini Fleming, Principal Investigator — University of Chicago Comprehensive Cancer Center
Locations (7):
- United States (4):
  - City of Hope Medical Center, Duarte, California
  - University of Southern California, Los Angeles, California
  - Decatur Memorial Hospital, Decatur, Illinois
  - Central Illinois Hematology Oncology Center, Springfield, Illinois
- Canada (3):
  - Juravinski Cancer Centre at Hamilton Health Sciences, Hamilton, Ontario
  - Cancer Centre of Southeastern Ontario at Kingston General Hospital, Kingston, Ontario
  - University Health Network-Princess Margaret Hospital, Toronto, Ontario

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study population consisted of patients at least 18 years old with advanced or recurrent carcinoma, or uterine carcinosarcoma. Both cohorts received a starting dose of 400 mg sorafenib orally twice daily on a continuous basis.
Pre-assignment Details: A Simon optimal two-stage design was used with objective response rate as the primary efficacy endpoint.
Groups:
- Carcinoma: Patients with advanced uterine carcinoma receive 400 mg oral sorafenib twice daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
- Carcinosarcoma: Patients with advanced uterine carcinosarcoma receive 400 mg oral sorafenib twice daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Carcinoma | Carcinosarcoma
Started | 40 | 16
Completed | 37 | 14
Not Completed | 3 | 2
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Adverse Event | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Carcinoma | Carcinosarcoma | Total
Number analyzed (Participants) | 40 | 16 | 56
Age, Customized [Median (Full Range); unit: years] | 64 [44 to 83] | 64 [40 to 87] | 64 [40 to 87]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 16 | 56
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  Non-Hispanic white | 29 | 10 | 39
  Hispanic | 4 | 1 | 5
  African-American | 2 | 3 | 5
  Asian | 5 | 2 | 7
Histology [Number; unit: participants]
  Adenocarcinoma (unspecified) | 12 | 0 | 12
  Serous | 3 | 0 | 3
  Clear cell | 1 | 0 | 1
  Endometrioid | 24 | 0 | 24
  Carcinosarcoma | 0 | 16 | 16

OUTCOME MEASURES:

1. Primary Outcome: Objective Overall Response Rate
Description: Response was defined using the Response Evaluation Criteria in Solid Tumors (RECIST, http://www.ncbi.nlm.nih.gov/pubmed/10655437#): Complete Response(CR), disappearance of all target lesions; Partial Response(PR), at least a 30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR)=CR+PR.
Time Frame: Up to 5 years
Measure: Number; unit: participants
Arm/Group | Carcinoma | Carcinosarcoma
Number analyzed (Participants) | 37 | 14
participants | 2 | 0

2. Secondary Outcome: Overall Survival
Description: Defined as the time from the first day of therapy to the date of death. If the patient was lost to follow-up, survival was censored on the last date the patient was known to be alive.
Time Frame: Up to 5 years
Measure: Median (95% Confidence Interval); unit: Month
Arm/Group | Carcinoma | Carcinosarcoma
Number analyzed (Participants) | 38 | 14
Month | 11.4 [6.9 to 17.7] | 5 [1.4 to 14]

3. Secondary Outcome: Progression Free Survival
Description: Defined as the time from the first day of treatment until the date PD(progressive disease) or death is first reported. Patients who died without a reported prior progression was considered to have progressed on the day of their death. Patients who did not progress was censored at the day of their last tumor assessment. According to RECIST, progressive disease(PD) is defined as at least a 20% increase in the sum of the longest diameter of target lesions.
Time Frame: Up to 5 years
Measure: Median (95% Confidence Interval); unit: Month
Arm/Group | Carcinoma | Carcinosarcoma
Number analyzed (Participants) | 38 | 14
Month | 3.2 [1.9 to 4] | 1.8 [1.4 to 3.5]

4. Secondary Outcome: Duration of Response
Description: Duration of response was measured from the time measurement criteria are met for CR(complete response)/PR(partial response), whichever was first recorded, until the first date that PD(progressive disease) was objectively documented. According to the RECIST: Complete Response(CR), disappearance of all target lesions; Partial Response(PR), at least a 30% decrease in the sum of the longest diameter of target lesions; progressive disease(PD), at least a 20% increase in the sum of the longest diameter of target lesions.
Time Frame: Up to 5 years
Measure: Mean (Full Range); unit: Month
Arm/Group | Carcinoma | Carcinosarcoma
Number analyzed (Participants) | 2 | 0
Month | 25 [10 to 40] |

ADVERSE EVENTS:
Arm/Group | Sorafenib
Serious Adverse Events (participants affected / at risk) | 11/56
Other Adverse Events (participants affected / at risk) | 56/56
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sorafenib (N=56)
Colitis, infectious (e.g., Clostridium difficile) (Infections and infestations) | 1
Death not associated with CTCAE term : Disease progression NOS (General disorders) | 2
Dehydration (Metabolism and nutrition disorders) | 1
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 1
Fatigue (asthenia, lethargy, malaise) (General disorders) | 1
Febrile neutropenia (fever of unknown origin without clinically or microbiologically documented infe (Blood and lymphatic system disorders) | 1
Fistula, GI : Colon/cecum/appendix (Gastrointestinal disorders) | 1
Fistula, GU : Vagina (Reproductive system and breast disorders) | 1
Hemorrhage, GI : Esophagus (Gastrointestinal disorders) | 1
Hemorrhage, GI : Lower GI NOS (Gastrointestinal disorders) | 1
Hemorrhage, GU : Bladder (Renal and urinary disorders) | 1
Hemorrhage, GU : Ureter (Renal and urinary disorders) | 1
Hypertension (Vascular disorders) | 1
Infection with unknown ANC : Bladder (urinary) (Infections and infestations) | 1
Infection with unknown ANC : Lung (pneumonia) (Infections and infestations) | 2
Infection with unknown ANC : Urinary tract NOS (Infections and infestations) | 1
Muscle weakness, generalized or specific area (not due to neuropathy) (Musculoskeletal and connective tissue disorders) | 1
Pain : Abdomen NOS (Gastrointestinal disorders) | 1
Pain : Joint (Musculoskeletal and connective tissue disorders) | 1
Phosphate, serum-low (hypophosphatemia) (Metabolism and nutrition disorders) | 1
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 1
Thrombosis/embolism (vascular access-related) (Injury, poisoning and procedural complications) | 2
Thrombosis/thrombus/embolism (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sorafenib (N=56)
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 13
Alkaline phosphatase (Investigations) | 16
ALT, SGPT (serum glutamic pyruvic transaminase) (Investigations) | 13
Anorexia (Metabolism and nutrition disorders) | 25
AST, SGOT(serum glutamic oxaloacetic transaminase) (Investigations) | 18
Bicarbonate, serum-low (Investigations) | 5
Bilirubin (hyperbilirubinemia) (Investigations) | 4
Calcium, serum-high (hypercalcemia) (Metabolism and nutrition disorders) | 6
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 14
Constipation (Gastrointestinal disorders) | 16
Cough (Respiratory, thoracic and mediastinal disorders) | 9
Diarrhea (Gastrointestinal disorders) | 24
Dizziness (Nervous system disorders) | 4
Dry skin (Skin and subcutaneous tissue disorders) | 10
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 8
Edema: limb (General disorders) | 10
Fatigue (asthenia, lethargy, malaise) (General disorders) | 27
Fever (in the absence of neutropenia, where neutropenia is defined as ANC <1.0 x 10e9/L) (General disorders) | 6
Flatulence (Gastrointestinal disorders) | 4
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 10
Glucose, serum-low (hypoglycemia) (Metabolism and nutrition disorders) | 3
Hair loss/alopecia (scalp or body) (Skin and subcutaneous tissue disorders) | 16
Heartburn/dyspepsia (Gastrointestinal disorders) | 4
Hemoglobin (Blood and lymphatic system disorders) | 21
Hemorrhage, GI : Rectum (Gastrointestinal disorders) | 5
Hemorrhage, pulmonary/upper respiratory : Nose (Respiratory, thoracic and mediastinal disorders) | 3
Hemorrhage, pulmonary/upper respiratory : Respiratory tract NOS (Respiratory, thoracic and mediastinal disorders) | 3
Hot flashes/flushes (Vascular disorders) | 4
Hypertension (Vascular disorders) | 18
INR (International Normalized Ratio of prothrombin time) (Investigations) | 5
Insomnia (Psychiatric disorders) | 7
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 12
Lymphopenia (Investigations) | 14
Mood alteration : Anxiety (Psychiatric disorders) | 3
Mucositis/stomatitis (functional/symptomatic) : Oral cavity (Gastrointestinal disorders) | 13
Muscle weakness, generalized or specific area (not due to neuropathy) : Extraocular (Musculoskeletal and connective tissue disorders) | 5
Nausea (Gastrointestinal disorders) | 20
Neuropathy: sensory (Nervous system disorders) | 5
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 4
Pain : Larynx (Respiratory, thoracic and mediastinal disorders) | 4
Pain : Abdomen NOS (Gastrointestinal disorders) | 24
Pain : Back (Musculoskeletal and connective tissue disorders) | 11
Pain : Bone (Musculoskeletal and connective tissue disorders) | 3
Pain : Extremity-limb (Musculoskeletal and connective tissue disorders) | 5
Pain : Head/headache (Nervous system disorders) | 5
Pain : Joint (Musculoskeletal and connective tissue disorders) | 9
Pain : Muscle (Musculoskeletal and connective tissue disorders) | 9
Phosphate, serum-low (hypophosphatemia) (Metabolism and nutrition disorders) | 15
Platelets (Investigations) | 7
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 15
Proteinuria (Renal and urinary disorders) | 3
Pruritus/itching (Skin and subcutaneous tissue disorders) | 4
Rash/desquamation (Skin and subcutaneous tissue disorders) | 26
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 18
Rash: hand-foot skin reaction (Skin and subcutaneous tissue disorders) | 20
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 11
Supraventricular and nodal arrhythmia : Sinus tachycardia (Cardiac disorders) | 3
Sweating (diaphoresis) (Skin and subcutaneous tissue disorders) | 3
Urinary frequency/urgency (Respiratory, thoracic and mediastinal disorders) | 3
Voice changes/dysarthria (e.g., hoarseness, loss or alteration in voice, laryngitis) (Respiratory, thoracic and mediastinal disorders) | 3
Vomiting (Gastrointestinal disorders) | 12
Weight loss (Investigations) | 14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less